CLINICAL TRIAL: NCT02698722
Title: A Video Decision Support Tool to Assist Elderly Patients in ESRD Treatment Decision-making - A Pilot Randomized Control Trial
Brief Title: A Video Decision Support Tool to Assist Elderly Patients in ESRD Treatment Decision-making
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Angelo E. Volandes, MD, Internist, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2014P002432
Record Dates: First submitted 2016-02-22; First posted 2016-03-04 (Estimated); Last update posted 2019-10-07 (Actual); Status verified 2019-10

CONDITIONS: Chronic Kidney Disease; Decision-making
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): This group will receive verbal education about dialytic and non-dialytic therapies via a standardized script.
- Intervention (Experimental): This group will receive the intervention which is a 11.5 minute video about dialysis and non-dialytic therapies.
  Interventions: Other: End-stage renal disease treatment options

INTERVENTIONS:
Other: End-stage renal disease treatment options — This group will receive the intervention which is a 11.5 minute video about dialysis and non-dialytic therapies.
  Arms: Intervention

SUMMARY:
In the United States, it is estimated that there are approximately 630,000 patients who have ESRD with two-thirds of those patients subsequently receiving maintenance dialysis. Studies have demonstrated that the initiation and timing of dialysis for those with ESRD seem to vary widely regionally - confirming the uncertainty of the benefits of chronic dialysis in this population

Pre-dialysis education programs inform patients of all of their options allowing them to choose renal replacement therapy that is most consistent with their wishes. Recent evidence has supported using different methods of delivering education including videos to complement standard clinical care practices to promote informed decision making. This proposed study will serve to examine the efficacy of a dialysis modality video decision support tool to inform chronic kidney disease patients of different dialytic and non-dialytic therapies.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking during clinical encounters
* Stage 4 or 5 CKD (defined by the Chronic Kidney Disease Epidemiology Collaboration for estimation of GFR < 30 ml/min/1.73m2)

Exclusion Criteria:

* Known history of dementia
* Legally blind
* Listed for kidney transplant

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-07-19 (Actual); Primary Completion 2019-03-22 (Actual); Study Completion 2019-03-22 (Actual)

PRIMARY OUTCOMES:
Change in knowledge of end-stage renal disease treatments (hemodialysis vs. peritoneal dialysis vs. supportive care) via survey | Change in knowledge immediately pre and post intervention and at 12 weeks

SECONDARY OUTCOMES:
Change in preference for end-stage renal disease treatment (hemodialysis vs. peritoneal dialysis vs. supportive care) via survey | Change in preferences Immediately pre and post intervention and at 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Eneanya ND, Percy SG, Stallings TL, Wang W, Steele DJR, Germain MJ, Schell JO, Paasche-Orlow MK, Volandes AE. Use of a Supportive Kidney Care Video Decision Aid in Older Patients: A Randomized Controlled Trial. Am J Nephrol. 2020;51(9):736-744. doi: 10.1159/000509711. Epub 2020 Aug 13. PMID 32791499